CLINICAL TRIAL: NCT04754542
Title: Discontinuation of Disease Modifying Therapies (DMTs) in Multiple Sclerosis (MS): Extension of the DISCOMS Study
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: EMD Serono (Industry); National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Other Study IDs: 20-2772
Record Dates: First submitted 2021-02-02; First posted 2021-02-15 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis
Keywords: Discontinuation; MS; DMT; Medication; Extension
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discontinuation: This study is only observing participants that received an intervention from a previous study. Participants that were randomized to discontinue their disease modifying therapy (DMT) in the DISCOMS study and consent to this extension trial will remain in this arm for the extension.
- Continuation: This study is only observing participants that received an intervention from a previous study. Participants that were randomized to continue their disease modifying therapy (DMT) in the DISCOMS study and consent to this extension trial will remain in this arm for the extension.

SUMMARY:
The Main Hypothesis of this extension trial is that among those who have successfully discontinued their DMT as part of the DISCOMS trial (i.e. did not have a new MS relapse or brain MRI lesion) and remain off DMT after DISCOMS are at no greater risk of new or worsened MS disease activity compared to those who successfully continued their DMT as part of DISCOMS and remain on DMT, each assessed at least one year after termination of the primary DISCOMS study.

DETAILED DESCRIPTION:
This will be a non-randomized, rater-blinded pragmatic trial, which is an extension of the randomized discontinuation trial (RDT), DISCOMS. While RDTs have been done in cancer, and rheumatoid arthritis patients, the original DISCOMS protocol was the first such study in MS. Study sites will be limited to the top 10 recruiting sites from the DISCOMS study due to financial and cost-effectiveness issues. Those sites will have participants who have completed 18-24 months of the primary study. In practice, the vast majority, if not all, will have completed 24 months. The investigators will explicitly include any who have completed, including those who already have exceeded 12 additional months after completion of the primary trial. Individuals who have successfully completed (retained original drug assignment and did not meet the primary endpoint of DISCOMS) the primary DISCOMS trial and are willing to retain their original drug assignment after completion and for an additional 12 months will be offered entry into the extension. The only exception to that will be individuals who continued the original drug assignment during and after the primary trial, up to 24 months, but who then had a relapse, new MRI lesion, or other MS-related reason between months 24 and 36 which resulted in their change of medication assignment. These individuals can and should be included, and counted as "failing" during the extension trial completing the Kaplan-Meier event free survival curve critical to the original hypothesis. A total of up to 100 patients will be consented and enter the extension trial, regardless of assignment, on a first come first serve basis to avoid selection biases to the extent possible. The intent is to take the first 100 who fulfill criteria and agree to participate. The plan is for a 50/50 distribution, but there may not be exactly 50 in each group. As of September 1, 2020, 102 had completed participation of the primary 24-month study, and information as to DMT use after finishing 2-years participation in DISCOMS was available for 46/102, 23 in each group (see Table 1 below). Notably, in the Discontinue group, 87% remained off DMT while only 61% in the Continue group remained on a DMT (13/14 on the same DMT, one switching to an alternative). Overall 74% remained in the primary assignment grouping. If these ratios stay consistent as more finish DISCOMS, discontinuers will account for roughly 59% of the total enrolled in the extension trial. Also, of the 102 completers, 20 have also gone at least an additional 12 months since completion of DISCOMS, and these participants will be offered entry into the extension trial, should these participants otherwise fulfill criteria. There will be no placebo and no sham treatment.

The study procedures will be slightly different for those who are completing Month 24 of the primary trial and simply "rolling over" to extension on the same day, compared to those who already have completed the study. For those rolling over at Month 24, DISCOMS participants will be offered participation in the extension trial. If these participants agree to participate, these participants will do a second study visit at the Month 24 visit, which concurrently will be Time Zero (T0) for the extension. This will consist of obtaining informed consent and going through Inclusion/Exclusion criteria. All the data from Month 24 visit will comprise the baseline data for the extension. Current and past DISCOMS study participants will be identified and screened for eligibility. This may include individuals who already have surpassed a full year since last participation in the trial, so long as these participants continued their original group assignment after the completion of the primary study and for at least for one additional year, or until a relapse or new MRI lesion occurred, as determined in screening. These individuals will explicitly be included, upon verification of the defining event. Patients will be approached at their next study visit or by phone (if these participants already completed the original study) by the PI and/or a study coordinator about participating in the study. The local PI for the study will verify accuracy of meeting inclusion criteria, and screening and consent may take place in person or by electronic means. Participants must agree to have a single SOC, month 36 MRI done by their primary neurologist and have the results and the MRI disk sent to the study site, to be assessed by a blinded central reader as has been done during the primary trial. All research visits will be conducted at the same time as SOC visits when possible, or as separate visits if not possible or the patient receives SOC elsewhere. For those who have exceeded 30 months from onset in the primary trial, the P1 visit (a telephone call) will not occur. All patients will undergo the T1 visit at 36 months, or longer should these participants have already exceed 36 months from onset of their participation in the primary trial.

A thorough discussion of the trial, signing the informed consent form, and confirmation of inclusion/exclusion criteria will be completed during the baseline visit (T0). Consenting may be done in-person on paper or using e-consent. If utilizing e-consent, participants will be presented a consent form ahead of time, and upon signature in the REDCap system, participants will receive a pdf of what was 'signed' electronically via REDCap. A pdf will also be generated for study records. T0 may occur on the same day as T1 if the patient has already completed the main DISCOMS study and is within the window for the Month 36 visit. There will be one phone call (P1), conducted by the study coordinator, at 30 Months post-enrollment in the original DISCO MS trial. On this phone call, the participant will be asked about any new or ongoing adverse events, changes to medications, and any symptoms suggesting a potential relapse. If the participant joins the Extension study after the participant already passed 30 Months post-enrollment in the original DISCO MS trial, the participant will not do P1. Those who have already exceeded 30 months since starting the primary DISCOMS trial will have the equivalent of the phone assessment at the T0 visit. Participants will come in for 1 additional study visit: T1 at 36 Months post-enrollment in the original DISCO MS trial. During T1, patients will undergo a blinded EDSS exam and relapse assessment, vitals, complete an SDMT assessment, and will complete all PROs/comorbidities. All PROs/comorbidities may be completed on paper in person or remotely via the electronic platform within the visit window, based on site and patient needs. Participants will also undergo a standard of care MRI scan of the brain at T1, within 60 days before and 120 days after the study visit. Participants who have already exceeded 12 months from the end of the primary trial will still be recruited and simply do the T1 visit at their earliest convenience. The maximum window will be 30 months after completion of the primary study, or 54 months since starting DISCOMS. Participants should always be brought in as close to 36 months as possible. Some participants' final study visit for the original DISCO MS study will be at 18 Months. For these subjects, the P1 visit will occur 24 Months after enrollment in the original study, and T1 will occur 30 Months after enrollment in the original study.

All participants will undergo the T1 visit, which will include a formal, blinded relapse assessment by the Examining Physician (EDSS rater) in conjunction with the PI (see section E). Prior to enrollment, the enrolling physician will certify, based on their personal review of the prior MRI scans and/or reports which will include data from the 24 month primary DISCOMS trial, that the scans have been stable for a minimum of 4.5 years (review of minimum of two scans, although it could be more, separated by at least 4.5 years). MRI scans at T1, 36+ months after onset of participation in the primary trial, will be performed as per usual SOC, paid for by patient insurance, at whatever site is normally used by the patient (preferably the same scanner each time, and preferably the same scanner as the investigation site), and should be done on a MRI machine with magnet 1.5 Tesla or greater, with and without contrast. Gadolinium may be withheld at the discretion of the PI or request of the patient. The window for T1 MRIs will be 60 day before or 120 days after the T1 study visit, and will be analyzed by a central, board-certified, blinded neuro-radiologist for new activity compared to prior scans. All MRI scans will be read locally for safety and clinical purposes, and PIs will communicate any significant MS or non-MS findings to the primary neurologist (should the investigator not be the primary neurologist). Any new lesion documented on the T1 MRI scan will prompt delivery of a notice within 48 hours, to the PI, that the patient has achieved the endpoint of the study, with a description of relevant findings.

In the event of a suspected relapse, the patient will be instructed to contact their physician and the study coordinator at their local site within 48 hours of new symptoms and come in for an unscheduled visit and relapse evaluation within seven days of symptom onset. Use of corticosteroids will be at the discretion of the patient and the local PI or other physician. Use of systemic steroids to treat MS symptoms will be concluded to be a Protocol-defined relapse. As at scheduled visits, the determination of a relapse at an unscheduled visit will be made by the blinded EDSS examiner, who will perform the EDSS and only then receive information about recent clinical history.

ELIGIBILITY:
Inclusion Criteria:

* Participation in and completion of the DISCOMS trial (NCT# 03073603) for a minimum of 18 and maximum of 24 months (i.e., it is possible some will have been enrolled late enough in the primary study so as to not have completed the full 24 months).

  o Only include participants in the following study groups
  * Randomized to the discontinue group, stayed off their DMT throughout and after the trial
  * Randomized to the continue group, continuously* stayed on their DMT throughout and after the trial
* Must be willing to continue in their previously-assigned treatment group for the entire, additional 12-Month follow-up period. For those in the continue group, the participant may have switched to a generic or biosimilar version of their medication, or to a different approved medication, if due to intolerance, convenience or insurance mandates, but NOT if due to having new or worsening MS disease activity.
* RRMS, SPMS, or PPMS by McDonald 2010 criteria. Patients will be defined by subtype based on 2013 updated phenotypic criteria. Progression of MS will be defined by the local principal investigator either prospectively with an EDSS change of at least 1.0 points over the last two years, or retrospectively, with any significant change in motor function over at least one year, unrelated to relapse.
* During the primary DISCOMS study, no evidence of recent new inflammatory disease activity (inactive by the Lublin criteria). Pseudorelapses due to infection, fever, or other stressors as deemed by the local PI will NOT be excluded. Those who have already successfully completed the primary DISCOMS study without having a new relapse or MRI scan change, but who have a relapse or scan change AFTER ending participation in DISCOMS but before entering the extension ARE eligible and will be recruited, i.e. we do not wish to undercount new activity that occurs after exiting DISCOMS.
* Provides informed consent to continue in the extension trial.
* Willing to follow the protocol.
* Able to undergo a brain MRI without anesthesia, as part of routine care (i.e. paid for by their insurance).

  * Continuously will be defined as no less than 75% of all prescribed doses, with no time of greater than four weeks from last intended dose to have missed a dose (8 weeks for natalizumab, i.e. one missed dose).

Exclusion Criteria:

* During original DISCOMS trial participant was randomized to the discontinue group, but then either re-started their DMT during the trial (study-defined 'treatment withdrawal), or wishes to restart their DMT after completing original DISCOMS study. Conversely, also excluded are those who completed the primary trial in the continue group and then discontinued, or wishes to discontinue, after completion of the primary study.
* Any MS relapse or new MRI scan lesion (3 mm or larger) during the primary DISCOMS trial, with relapse determined by the blinded examiner and MRI lesion determined by the blinded MRI reader.
* Significant (as defined by the PI) intolerance of presently-used DMT, if taking a DMT
* The following must not have occurred during the original DISCO MS study or since completing the study:

  * Use of any non-FDA-approved DMT
  * More than two courses of acute, systemic (IV or oral). Course is defined as three or more days continuously, and not to exceed 14 days. No use of chronic, systemic steroids, defined as 15 or more days. Any use of steroids to treat MS relapse, possible relapse, or pseudo-relapse is excluded. Inhaled or topical steroids for non-MS are not exclusionary.
  * Use of alemtuzumab, mitoxantrone, cyclophosphamide, methotrexate, cyclosporine, rituximab, or cladribine.
  * Use of any experimental agent used as a DMT for MS
  * Cancers other than basal cell skin cancers
* Other significant medical or psychiatric illness, if uncontrolled. Examples: uncontrolled hypertension, uncontrolled diabetes, uncontrolled asthma, uncontrolled depression.
* Unable to give informed consent or follow the protocol.
* Unable to undergo brain MRI.
* History of other chronic neurological illnesses that might mimic MS with chronic or intermittent symptoms (i.e. ALS, myasthenia gravis, chronic neuropathy, etc.).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is limited to subjects that are currently participating in or have completed the DISCOMS trial (NCT# 03073603). Only subjects that remained in their original treatment arm throughout the trial as well as those that remained in their treatment arm after their participation was completed will qualify. Participants in the DISCOMS trial that experienced a relapse during the study will not qualify for the extension.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Corboy, MD, Principal Investigator — University of Colorado, Denver
Locations (10):
- United States (10):
  - University of Colorado Denver, Aurora, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - New York University, New York, New York
  - Mount Sinai, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Swedish, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study population is limited to subjects that are currently participating in or have completed the DISCOMS trial (NCT# 03073603). Only subjects that remained in their original treatment arm throughout the trial as well as those that remained in their treatment arm after their participation was completed will qualify. Participants in the DISCOMS trial that experienced a relapse during the study will not qualify for the extension.
Period: Overall Study
Arm/Group | Continuation | Discontinuation
Started | 31 | 45
Completed | 30 | 44
Not Completed | 1 | 1
Not completed — Subject enrolled in error; did not meet eligibility criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Discontinuation | Continuation | Total
Number analyzed (Participants) | 44 | 30 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (4.7) | 61 (4.4) | 62.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 25 | 63
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 3 | 4 | 7
  White | 41 | 26 | 67
Region of Enrollment [Number; unit: participants]
  United States | 44 | 30 | 76
MS Phenotype [Count of Participants; unit: Participants]
  Relapsing-Remitting | 40 | 29 | 69
  Secondary Progressive | 4 | 1 | 5
Time since first onset of symptoms related to MS [Mean (Standard Deviation); unit: years] | 23.7 (9.5) | 17.1 (7.4) | 21.0 (9.3)
Time since last documented relapse [Mean (Standard Deviation); unit: years] | 14.5 (6) | 11.5 (5.1) | 13.3 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Off Drug That Have New Inflammatory Disease Compared to Those on Drug.
Description: As inflammatory disease activity may be manifested clinically as a relapse, or radiographically as a new MRI lesion, we have chosen a combined primary outcome measure.
Time Frame: Month 36 visit. The Month 36 visit was the extension study's only visit, which occurred 36 months after randomization in the original DISCOMS study (NCT03073603).
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation | Continuation
Number analyzed (Participants) | 44 | 30
Participants | 2 | 1
Statistical Analysis 1: Comparison: Discontinuation vs Continuation; We tested the null hypothesis of inferiority with the proportion of disease events (i.e., new MS relapse and/or MRI brain lesion) for the drug discontinuation group being 8% greater than the proportion for the drug continuation group under the alternative that the two rates are equal; Test type: Non-Inferiority — We performed a non-inferiority test for the proportions of the drug continuation and drug discontinuation arms experiencing a new MS relapse and/or MRI Brain Lesion over the course of the study duration. The non-inferiority margin used was 8%; p = 0.124, Exact binomial test; Exact binomial test fr difference in two proportions; Difference in proportion = 0.0121, 95% CI 2-sided [-0.1321 to 0.1287]

2. Secondary Outcome: Compare the Change in Disability Using the EDSS Over the Duration of the Trial in Those Who Were Able to Maintain Their Treatment Assignment Without Inflammatory Activity.
Description: The Expanded Disability Status Scale (EDSS) is a commonly used assessment that allows clinicians to objectively measure changes in a patient's symptoms by using unbiased raters. This assessment will be collected at all time-points and will be used to measure changes in patients' symptoms over the course of the study and will be used to help define 'relapse', i.e. will require a change on examination. Possible scores range from 0 to 10, with higher scores indicating a worse outcome (i.e. more severe disability)
  The change between baseline of the original DISCOMS study (NCT03073603) and Month 36 is reported.
Time Frame: Baseline of the original DISCOMS study (NCT03073603) and Month 36. The Month 36 visit was the extension study's only visit, which occurred 36 months after randomization in the original DISCOMS study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 28 | 44
score on a scale | 0 (0.82) | 0.10 (0.94)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.639, t-test, 2 sided

3. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Upper Extremity Function
Description: The Neuro-QOL Adult PRO short form measures are self-reported measures of overall quality of life and functioning. The Neuro-Qol short form scales consist of 5-9 single scale item scales. Raw scores are then converted to a standardized score with mean 50 and standard deviation 10. The Neuro-QoL short forms used in this study with higher scores representing better outcomes are: Upper Extremity Function, Lower Extremity Function, Cognitive -- General Concerns, Cognitive -- Executive Function, Communication, Positive Affect and Well-Being, Satisfaction with Social Roles and Activities, and Ability to Participate in Social Roles and Activities. The short forms used with lower scores representing better outcomes are: Fatigue, Sleep Disturbance, Anxiety, Depression, and Emotional-Behavioral Dyscontrol. The change between baseline of the original DISCOMS study (NCT03073603) and Month 36 is reported.
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | 0.2 (5.1) | 0.1 (4.3)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.964, t-test, 2 sided

4. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Lower Extremity Function
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | 0.4 (7) | -0.6 (5)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.819, t-test, 2 sided

5. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Fatigue
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | -0.2 (5.7) | 0.6 (5.1)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.515, t-test, 2 sided

6. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Sleep Disturbance
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | -0.5 (5.8) | 0.6 (5.5)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.388, t-test, 2 sided

7. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- General Concerns
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | 0.5 (3.7) | 2.3 (6.5)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.183, t-test, 2 sided

8. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Executive Function
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | 1 (5.8) | -0.2 (6.8)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.414, t-test, 2 sided

9. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Communication
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 28 | 43
units on a scale | -0.1 (2.1) | -0.1 (2.3)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.998, t-test, 2 sided

10. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Anxiety
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | -0.2 (4.8) | 1.3 (7.1)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.320, t-test, 2 sided

11. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Depression
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | -1.2 (5.2) | 1.3 (5.4)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.061, t-test, 2 sided

12. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Positive Affect and Well-Being
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | 2.5 (6.4) | -0.8 (6.2)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.032, t-test, 2 sided

13. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Emotional-Behavioral Dyscontrol
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | 0.7 (7.4) | -0.3 (6.5)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.514, t-test, 2 sided

14. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Satisfaction With Social Roles and Activities
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | 0.9 (4.5) | -2.3 (6.2)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.017, t-test, 2 sided

15. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - NeuroQoL Short Form Scores -- Ability to Participate in Social Roles and Activities
Description: as for outcome 3
Time Frame: as for outcome 2
Population: Subjects missing Neuro-QoL at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 43
units on a scale | -1.1 (8.3) | -4.3 (9.6)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.155, t-test, 2 sided

16. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - SymptoMScreen
Description: SymptoMScreen is a rapid assessment tool that allows the patient to self-report across multiple neurological domains (mobility, hand function, spasticity, pain, sensory, bladder, fatigue, vision, dizziness, cognition, depression, and anxiety). This scale is a user friendly, single page validated measure that allows for quick assessment of multiple symptoms. Single item scores are rated as 0-6 with higher numbers representing increased limitations and symptom severity. Composite score is calculated by summing the single item scores with total score ranges from 0 to 72.
  The change between baseline of the original DISCOMS study (NCT03073603) and Month 36 is reported.
Time Frame: as for outcome 2
Population: Subjects missing SymptoMScreen at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 30 | 44
units on a scale | 0 (0.5) | 0.1 (0.5)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.358, t-test, 2 sided

17. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - Patient Determined Disease Steps (PDDS)
Description: The Patient-Determined Disease Steps (PDDS) is a PRO version of the clinician-reported Extended Disability Status Scale (EDSS) which hones the stages of cane use and thus is more responsive to mid-range disability changes. This tool asks the patient to characterize level of disability into one of nine steps (0=normal, 1=mild disability, 2=moderate disability, 3=gait disability, 4=early cane, 5=late cane, 6=bilateral support, 7=wheelchair scooter, 8=bedridden). The PDDS will be used to characterize (and to control for) disability in both study groups at all study time points.
  The change between baseline of the original DISCOMS study (NCT03073603) and Month 36 is reported.
Time Frame: as for outcome 2
Population: Subjects missing PDDS at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 44
units on a scale | -0.1 (0.8) | 0.3 (1.1)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.151, t-test, 2 sided

18. Other Pre Specified Outcome: Patient Reported Outcomes (PROs) - Change in Symbol Digit Modalities Test (SDMT)
Description: The SDMT measures patient attention, concentration, and speed of information processing and has been validated for discriminating patients from controls even when it was administered each month over six months. It is relatively simple to administer and only takes a few minutes to complete. Possible scores range from 0 to 110, with higher scores indicating a better outcome.
  The change between baseline of the original DISCOMS study (NCT03073603) and Month 36 is reported.
Time Frame: as for outcome 2
Population: Subjects missing SDMT at either DISCOMS baseline or at Month 36 were excluded from this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 28 | 43
units on a scale | 4.8 (10.2) | 1.4 (7.9)
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.123, t-test, 2 sided

19. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - Multiple Sclerosis Impact Scale (MSIS-29) -- Psychological Impact
Description: Since Neuro-QoL short form doesn't have the ability to provide an overall quality of life calculation, the study team added MSIS-29, which is an acceptable, reliable, and valid method for recording quality of life in MS patients. The Multiple Sclerosis Impact Scale (MSIS-29) will be collected to assess changes in quality of life from the patient's perspective. The MSIS has 29 questions. Each question asks the participant to rank how impacted they are in a certain aspect of their life. The options are 1 through 4. 1 indicates not at all impacted while 4 indicates extremely impacted. The lower the final score, the less impacted the participant is overall. Scores on the physical impact scale range from 20-80 and from 9-36 on the psychological impact scale. We will compare the proportion in each group who have had a change of 7.5 points or more (considered a clinically meaningful change).
  The change between baseline of the original DISCOMS study (NCT03073603) and Month 36 is reported.
Time Frame: as for outcome 2
Population: Subjects missing MSIS-29 at either baseline or at Month 36 were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 44
Participants
  Significant change | 11 | 19
  No significant change | 18 | 25
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.656, Chi-squared

20. Other Pre Specified Outcome: Change in Patient Reported Outcomes (PROs) - Multiple Sclerosis Impact Scale (MSIS-29) -- Physical Impact
Description: as for outcome 19
Time Frame: as for outcome 2
Population: Subjects missing MSIS-29 at either baseline or at Month 36 were excluded from this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 29 | 44
Participants
  Significant change | 11 | 16
  No significant change | 18 | 28
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.892, Chi-squared

21. Other Pre Specified Outcome: Patient Reported Outcomes (PROs) - Treatment Satisfaction Questions
Description: This was developed for qualitative and exploratory purposes. These questions will provide insight into patient satisfaction in regards to the disease modifying therapy (DMT) they are using at baseline, versus their ongoing satisfaction with their study care plan (on a DMT v. not on a DMT). Patients were asked, "How Satisfied Are You with Your Present DMT or Lack of DMT?", and could respond on a five-point scale as Highly unsatisfied, Unsatisfied, Neutral, Satisfied, or Highly Satisfied.
Time Frame: Month 36 visit. The Month 36 visit was the extension study's only visit, which occurred 36 months after randomization in the original DISCOMS study.
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation | Discontinuation
Number analyzed (Participants) | 28 | 40
Participants
  Very dissatisfied | 3 | 5
  Dissatisfied | 0 | 0
  Neutral | 7 | 0
  Satisfied | 4 | 6
  Very satisfied | 14 | 29
Statistical Analysis 1: Comparison: Continuation vs Discontinuation; Test type: Superiority; p = 0.063, Mantel Haenszel; Cochran-Mantel-Haenszel chi-square test for ordinal-nominal association was used

22. Other Pre Specified Outcome: Patient Reported Outcomes (PROs) - Treatment Decision Questions (Continuation Group)
Description: These questions were also developed for exploratory purposes to gain insight on the MS DMT treatment decisions at the conclusion of the study and to better understand recruitment and retention, for patients who were randomized to either staying on or going off their DMT.
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Continuation
Number analyzed (Participants) | 29
Participants
  Stop my DMT | 4
  Continue my current DMT | 25
  Switch to a new DMT | 0

23. Other Pre Specified Outcome: Patient Reported Outcomes (PROs) - Treatment Decision Questions (Discontinuation Group)
Description: as for outcome 22
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation
Number analyzed (Participants) | 42
Participants
  Stay off my DMT | 42
  Restart a prior DMT | 0
  Restart a new DMT | 0

ADVERSE EVENTS:
Time Frame: Baseline to end of study (18 months)
Description: All adverse events and serious adverse events are reported.
Arm/Group | Continuation | Discontinuation
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/44
Other Adverse Events (participants affected / at risk) | 4/30 | 3/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuation (N=30) | Discontinuation (N=44)
Overactive and neurogenic bladder (Renal and urinary disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuation (N=30) | Discontinuation (N=44)
Increased arthritis pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pelvic organ prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
chills, fatigue and body aches following COVID-19 vaccine (Immune system disorders) | 1 (1) | 0 (0)
trigeminal neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
COVID-19 infection (Infections and infestations) | 1 (1) | 0 (0)
bronchitis (Infections and infestations) | 0 (0) | 1 (1)
ostopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT04754542/Prot_SAP_000.pdf